CLINICAL TRIAL: NCT00242671
Title: The Efficacy of Isocapnic Hyperpnoea to Accelerate Recovery After General Anesthesia With Sevoflurane.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Rita Katznelson, Toronto General Hospital, University Health Network
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UHN REB 05-0299-AE
Record Dates: First submitted 2005-10-18; First posted 2005-10-20 (Estimated); Last update posted 2010-08-05 (Estimated); Status verified 2006-09

CONDITIONS: Anesthesia
Keywords: general anesthesia, hyperventilation, carbon dioxide, isocapnic hyperponea
MeSH Terms: conditions — Hyperventilation

INTERVENTIONS:
Procedure: Isocapnic Hyperponea

SUMMARY:
The twilight phase between being asleep and awake during recovery from anesthesia is a precarious time fraught with risks to the post-operative patient. Hyperventilation accelerates the elimination of inhaled anesthetics but reduces their CO2 blood concentrations which delays their resumption of spontaneous breathing. We previously showed that our method of hyperventilation without affecting the CO2 concentration--which we call IH--accelerates the rate of emergence from anesthesia with isoflurane. In this study we will study the effect of IH on the rate of emergence from Sevoflurane anesthesia.

ELIGIBILITY:
Inclusion criteria:

1. Elective gynecological procedure
2. ASA I-III
3. Age 18-80 years
4. Signed informed consent

Exclusion criteria:

1. ASA IV
2. Patients with contra-indications to Sevoflurane anesthesia or other anesthetics included in the protocol
3. Active smoking, asthma or other history of hyper-reactive airway disease
4. History of chronic obstructive lung disease limiting exercise
5. History of angina, previous myocardial infarction, valvular heart disease, or heart surgery
6. Presence of heart murmurs or neck bruits
7. ECT abnormalities including atrial fibrillation, prolonged P-R interval, prolonged Q-T interval, presence of Q waves in inferior, anterior or lateral leads, criteria for left ventricular hypertrophy, T-wave abnormalities,
8. History of difficult airway access
9. Pulmonary hypertension and/or right ventricle dysfunction
10. History of bulous emphysema, and/or spontaneous pneumothorax
11. History of alcohol or drugs abuse
12. Known history of psychiatric illness and/or medications
13. Patients that required postoperative mechanical ventilation for any reason

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2005-10; Primary Completion 2008-08 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Time to recovery from anesthesia as indicated by time to extubation and rate of change of BIS score

SECONDARY OUTCOMES:
Quality of recovery in the recovery room as indicated by the level of consciousness, incidence of nausea, vomiting, shivering and other phenomena occuring during recovery

CONTACTS AND LOCATIONS:
Overall Officials: Rita Katznelson, MD, Principal Investigator — Toronto General Hospital, University Health Network
Locations (1):
- Toronto General Hospital, University Health Network, Toronto, Ontario, Canada